CLINICAL TRIAL: NCT00644189
Title: A Phase II Study of Oral Clofarabine in Patients With Relapsed/Refractory Non-Hodgkin Lymphoma
Brief Title: Oral Clofarabine for Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-401
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma; Low Grade B-cell Lymphoma, Not Otherwise Specified; Diffuse Large B-cell Lymphoma; Peripheral T-cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large-cell Lymphoma
Keywords: clofarabine; Clolar; lymphoma; NHL; oral chemotherapy
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clofarabine (Other): Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
  Other Names: Clolar

SUMMARY:
Oral clofarabine is related to two intravenous chemotherapy drugs used for this disease and works in two different ways. It affects the development of new cancer cells by blocking two enzymes that cancer cells need to reproduce. When these enzymes are blocked, the cancer call can no longer prepare the DNA needed to make new cells. Clofarabine also encourages existing cancer cells to die by disturbing components within the cancer cell. This causes the release of a substance that is fatal to the cell.

This trial studies the efficacy of oral clofarabine in the treatment of relapsed non-Hodgkin lymphomas.

DETAILED DESCRIPTION:
* Each treatment cycle lasts four weeks during which time the participant will be taking study drug for the first three weeks only. Participants will be supplied with a study medication-dosing calendar for each treatment cycle.
* Clofarabine is a tablet that will be taken orally in the morning once daily on days 1 through 21 of each 28-day cycle. Participants can receive up to a total of 6 cycles if they do not experience any unacceptable side effects and if their cancer does not get worse.
* The following tests and procedures will be performed at specified intervals through out the treatment period: blood tests, physical examinations, vital signs, radiological exams and urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory NHL that includes: follicular lymphoma of any grade; marginal zone lymphoma; small lymphocytic lymphoma/chronic lymphocytic leukemia; mantle cell lymphoma; lymphoplasmacytic lymphoma; low-grade B-cell lymphoma not otherwise specified; diffuse large B-cell lymphoma, anaplastic large cell lymphoma, peripheral T-cell lymphoma, angioimmunoblastic T-cell lymphoma.
* One or more prior line of chemotherapy, immunotherapy, or radioimmunotherapy.
* Measurable disease on cross sectional imaging of at least 2cm.
* ECOG Performance Status 0-2
* 18 years of age or older
* Life expectancy of greater than 3 months
* Normal organ and marrow function as outlined in the protocol
* Must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Patients who have had chemotherapy, rituximab, or radiotherapy within 4 weeks, or radioimmunotherapy within 8 weeks prior to entering the study
* Receiving any other investigational agent
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Clofarabine
* Systemic fungal, bacterial, viral, or other infection not controlled
* Pregnant or lactating
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for over one year
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior allogeneic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine 1 mg; Clofarabine 2 mg; Clofarabine 4 mg; Clofarabine: 3 mg: Clofarabine: Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
Period: Phase I
Arm/Group | Clofarabine 1 mg | Clofarabine 2 mg | Clofarabine 4 mg | Clofarabine: 3 mg
Started | 3 | 3 | 6 | 18
Completed | 3 | 3 | 6 | 18
Not Completed | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Clofarabine 1 mg | Clofarabine 2 mg | Clofarabine 4 mg | Clofarabine: 3 mg
Started | 0 (All phase I participants were included in the 3mg Phase II dose group) | 0 (All phase I participants were included in the 3mg Phase II dose group) | 0 (All phase I participants were included in the 3mg Phase II dose group) | 50 (Additional participants were added to the phase I sample at the phase II 3mg dose level)
Completed All 6 Cycles of Treatment | 0 | 0 | 0 | 19
Completed | 0 | 0 | 0 | 50
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase I participants
Groups:
- Clofarabine Phase I: Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
  Clofarabine: Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
Arm/Group | Clofarabine Phase I
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30
Number of prior regimens [Median (Full Range); unit: number of prior regimens] | 1 [1 to 7]
Histologies [Count of Participants; unit: Participants]
  follicular lymphoma (FL) | 7
  small lymphocytic lymphoma (SLL) | 6
  diffuse large B-cell lymphoma (DLBCL) | 3
  marginal zone lymphoma (MZL) | 7
  mantle cell lymphoma (MCL) | 6
  T-cell lymphoma (TCL) | 0
  lymphoplasmacytic lymphoma (LPL) | 1

OUTCOME MEASURES:

1. Primary Outcome: All Phase I-II Participants: Overall Response Rate (ORR)
Description: Determine the efficacy of oral clofarabine (any of the 4 dose levels: 1mg, 2mg, 4mg, and 3mg) in all phase I-II trial patients with relapsed/refractory non-Hodgkin lymphomas.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: after at most 6 28-day cycles
Population: all participants from phase I-II trial who are treated with any of the 4 dose levels of oral clofarabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I-II: Clofarabine: Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
Arm/Group | Phase I-II
Number analyzed (Participants) | 50
percentage of participants | 28 [16 to 42]

2. Primary Outcome: Phase I Participants Only: Overall Response Rate (ORR)
Description: Determine the efficacy of oral clofarabine (any of the 4 dose levels: 1mg, 2mg, 4mg, and 3mg) in all phase I trial patients with relapsed/refractory non-Hodgkin lymphomas.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: after at most 6 28-day cycles
Population: Phase I participants only
Measure: Mean (90% Confidence Interval); unit: percentage of participants
Groups:
- Phase I: Clofarabine: Taken orally once a day (in the AM) on days 1 through 21 of a 28-day cycle for a maximum of 6 cycles.
Arm/Group | Phase I
Number analyzed (Participants) | 30
percentage of participants | 47 [31 to 63]

3. Secondary Outcome: Phase I-II Participants Treated at the RP2D (3mg): Overall Response Rate (ORR)
Description: To determine the efficacy of oral clofarabine (3mg) in patients with relapsed/refractory non-Hodgkin lymphoma. The 3mg dose was declared the recommended phase 2 dose (RP2D) from phase I.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: after at most 6 28-day cycles
Population: only participants from phase I-II trial who were treated at the RP2D (3mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 36
percentage of participants | 28 [14 to 45]

4. Secondary Outcome: All Phase I-II Participants: Progression-free Survival (PFS)
Description: Determine the progression-free survival rate among all phase I-II trial participants who are treated with any of the 4 dose levels of oral clofarabine (1mg, 2mg, 4mg, or 3mg).
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: at 1 and 2 years
Population: all participants from phase I-II trial who are treated with any of the 4 dose levels of oral clofarabine
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Clofarabine
Number analyzed (Participants) | 50
percentage of patients
  1-year PFS | 32 [20 to 45]
  2-year PFS | 16 [7.5 to 27]

5. Secondary Outcome: All Phase I-II Participants: Overall Survival (OS)
Description: Determine the overall survival rate among all phase I-II trial participants who are treated with any of the 4 dose levels of oral clofarabine (1mg, 2mg, 4mg, or 3mg)
Time Frame: 3 years
Population: all participants from phase I-II trial who are treated with any of the 4 dose levels of oral clofarabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 50
percentage of participants | 58 [43 to 71]

6. Secondary Outcome: All Phase I-II Participants: Safety
Description: Grade 3-4 toxicities among all phase I-II trial participants who are treated with any of the 4 dose levels of oral clofarabine (1mg, 2mg, 4mg, or 3mg)
Time Frame: during 6 28-day cycles and 90 days out
Population: all phase I-II trial participants who are treated with any of the 4 dose levels of oral clofarabine
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 50
Participants
  Any grade 3-4 toxicity | 29
  Leukopenia and neutropenia | 24
  Thrombocytopenia | 15
  Anemia | 7
  Fatigue | 3

7. Secondary Outcome: Phase I Participants Treated at the RP2D (3mg): Overall Response Rate (ORR)
Description: as for outcome 3
Time Frame: after at most 6 28-day cycles
Population: Phase I participants only who were treated at the RP2D (3mg)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I
Number analyzed (Participants) | 16
Participants
  Complete Response (CR) | 5
  Partial Response (PR) | 4
  Stable Disease (SD) or Progressive Disease (PD) | 7

8. Secondary Outcome: Phase I Participants: Progression-free Survival (PFS)
Description: Determine the progression-free survival rate among all phase I trial participants who are treated with any of the 4 dose levels of oral clofarabine (1mg, 2mg, 4mg, or 3mg).
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: at 17 months
Population: Phase I participants only
Measure: Mean (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I
Number analyzed (Participants) | 30
percentage of participants | 34 [17 to 51]

9. Secondary Outcome: All Phase I Participants: Overall Survival (OS)
Description: Determine the overall survival rate among all phase I trial participants who are treated with any of the 4 dose levels of oral clofarabine (1mg, 2mg, 4mg, or 3mg)
Time Frame: at 17 months
Population: Phase I participants only
Measure: Mean (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I
Number analyzed (Participants) | 30
percentage of participants | 75 [62 to 89]

10. Secondary Outcome: Phase I Participants: Safety
Description: Grade 2-4 toxicities and grade 3-4 infections among all phase I trial participants who are treated with any of the 4 dose levels of oral clofarabine (1mg, 2mg, 4mg, or 3mg)
Time Frame: during 6 28-day cycles and 90 days out
Population: Phase I participants only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I
Number analyzed (Participants) | 30
Participants
  Anemia | 19
  Neutropenia | 18
  Thrombocytopenia | 9
  Fatigue | 8
  Neutropenic fever | 1
  Grade 3-4 infections | 3
  Any grade 3-4 toxicity | 20

ADVERSE EVENTS:
Arm/Group | Clofarabine
Serious Adverse Events (participants affected / at risk) | 15/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=50)
Anemia (Blood and lymphatic system disorders) | 5 (6)
CNS Cerebrovascular Ischemia (Nervous system disorders) | 1 (1)
CNS Hemorrhage (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Death (due to disease Progression) (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Kidney Failure (Renal and urinary disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Pain - Left Flank (General disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Petechia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
suspected GI Bleed (Gastrointestinal disorders) | 1 (1)
Suspected respiratory tract infection (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7)
Weakness in legs (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=50)
Chills (General disorders) | 50 (255)
Ascites (Gastrointestinal disorders) | 50 (254)
Platelets (Blood and lymphatic system disorders) | 50 (253)
Febrile neutropenia (Blood and lymphatic system disorders) | 50 (253)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 50 (253)
Nausea (Gastrointestinal disorders) | 50 (252)
Vomiting (Gastrointestinal disorders) | 50 (252)
Leukocytosis (Blood and lymphatic system disorders) | 50 (252)
Head/headache (General disorders) | 50 (252)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 50 (244)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 12 (27)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 11 (24)
Brachial plexopathy (Nervous system disorders) | 11 (16)
Constipation (Gastrointestinal disorders) | 11 (15)
Hypokalemia (Metabolism and nutrition disorders) | 10 (32)
AST, SGOT (Metabolism and nutrition disorders) | 10 (17)
Dehydration (Metabolism and nutrition disorders) | 8 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (14)
Movements involuntary (Nervous system disorders) | 7 (17)
Back, pain (General disorders) | 7 (12)
Joint, pain (General disorders) | 7 (10)
Abdomen, pain (General disorders) | 7 (9)
Chemoradiation dermatitis (Skin and subcutaneous tissue disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 6 (9)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (16)
Edema limb (Blood and lymphatic system disorders) | 5 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (11)
Allergic rhinitis (Immune system disorders) | 5 (9)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (9)
Hypernatremia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 4 (13)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (9)
Insomnia (General disorders) | 4 (8)
Anorexia (Gastrointestinal disorders) | 4 (7)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 4 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Fatigue (General disorders) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (7)
Pelvic, pain (General disorders) | 3 (6)
Infection Gr0-2 neut, skin (Infections and infestations) | 3 (5)
Cardiac-other (Cardiac disorders) | 3 (4)
Fever w/o neutropenia (General disorders) | 3 (4)
Weight loss (General disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Pain-other (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes